CLINICAL TRIAL: NCT06122428
Title: Modified Sodium Hyaluronate Conjugated to Riboflavin (HAr® 0.1%) as Lubricant Eyedrops in the Treatment of Dry Eye
Brief Title: Efficacy of Riboflavin-Enhanced Hyaluronic Acid Eye Drops in Treating Dry Eye Disease
Status: Completed | Type: Observational
Sponsor: University of Naples (Other)
Responsible Party: Principal Investigator, Luca D'Andrea, Prinicipal investigator, Federico II University
Other Study IDs: CIT_001
Record Dates: First submitted 2023-10-12; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye Disease
Keywords: dry eye disease; ribohyal; ocular surface; tear check
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group X: Ribohyal Group: Composed of 16 eyes (right or left) assigned for the use of modified hyaluronic acid, HAr® 0.1%, covalently linked to Riboflavin
  Interventions: Drug: modified hyaluronic acid 0.1% covalently linked to Riboflavin
- Group Y: (Control Group): Composed of 16 eyes (right or left) assigned for the use of HA 0.1% alone
  Interventions: Drug: hyaluronic acid 0.1%

INTERVENTIONS:
Drug: modified hyaluronic acid 0.1% covalently linked to Riboflavin — The patients used the eye drops no less than 3 times a day or no more than 6 times a day, according to their needs. They reported the instillation frequency (3/4 or 5/6 times per day) on the provided document
  Groups: Group X: Ribohyal Group
Drug: hyaluronic acid 0.1% — The patients used the eye drops no less than 3 times a day or no more than 6 times a day, according to their needs. They reported the instillation frequency (3/4 or 5/6 times per day) on the provided document
  Groups: Group Y: (Control Group)

SUMMARY:
The goal of this retrospective study is to evaluate the historical effectiveness of Riboflavin-Enhanced Hyaluronic Acid Eye Drops (HAr® 0.1%) in the treatment of Dry Eye Disease (DED) among patients. The product under investigation, Ribohyal®, had previously obtained certification and authorization from the relevant notified body for market sale (European patent n. 2228058)

The primary questions it aimed to address were:

* Did the use of Riboflavin-Enhanced Hyaluronic Acid Eye Drops result in a reduction of dry eye symptoms and an improvement in ocular comfort among patients with DED in a historical context?
* Was Riboflavin-Enhanced Hyaluronic Acid Eye Drops historically more effective in reducing photophobia and enhancing tear film stability when compared to standard treatment?

Participants in this retrospective analysis had historically:

* Used either Riboflavin-Enhanced Hyaluronic Acid Eye Drops or a standard hyaluronic acid eye drop, based on their assigned group.
* Historically reported their levels of ocular discomfort and photophobia at specified time points.
* Undergone historical clinical examinations to assess tear film stability and osmolarity.

Researchers conducted a retrospective analysis to compare the historical outcomes of the group using Riboflavin-Enhanced Hyaluronic Acid Eye Drops with the group using standard eye drops to determine if the former historically provided more significant improvements in dry eye symptoms and tear film stability.

DETAILED DESCRIPTION:
In this retrospective study, the investigators have examined the historical therapeutic efficacy of Riboflavin-Enhanced Hyaluronic Acid Eye Drops (HAr® 0.1%) in the treatment of Dry Eye Disease (DED), adhering to good clinical practice principles.

Participants were historically divided into two groups:

* Group X: received Riboflavin-Enhanced Hyaluronic Acid Eye Drops (HAr® 0.1%) (Ribohyal Group).
* Group Y: received standard HA 0.1% eye drops (Control Group).

The historical outcome measures included the retrospective assessments of osmolarity, Tear Break-Up Time (TBUT), corneal staining, Schirmer test, tear meniscus measurement, and Non-invasive Break-Up Time (NIBUT). The Ocular Surface Disease Index (OSDI) score was historically recorded at various time points.

ELIGIBILITY:
Inclusion criteria for patient selection included a dry eye history of at least three months, OSDI score ≥ 23, and positivity in at least one eye for one or more of the following diagnostic criteria:

* Tear Break-Up Time (TBUT) < 7 seconds
* Schirmer test I at 5 minutes < 10 mm
* Corneal and/or conjunctival fluorescein staining
* Tear osmolarity > 308 mOsm/L or a difference of at least 8 mOsm/L between both eyes.

Exclusion Criteria:

* Age below 18 years
* Severe ocular surface affections
* Unilateral dry eye syndrome
* Refractive surgery performed within the last six months
* Eye surgery performed within the last three months
* Previous herpetic keratitis
* Signs of active corneal infection
* Systemic or topical steroid therapy within the last 30 days
* Topical therapy within the last 14 days
* Inability to understand the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study enrolled 16 consecutive patients with bilateral mild to severe Dry Eye Disease (DED) at the University of Naples Federico II, Italy. These participants were selected based on specific eligibility criteria, as outlined in other sections of the study. The selection aimed to ensure that the study population adequately represented individuals experiencing DED.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy and safety of a new 0.1% sodium hyaluronate-riboflavin-conjugated (HAr®) artificial tear in treating ocular discomfort and improving tear film stability in patients with dry eye disease. | From enrollment to the end of treatment at 8 weeks
  Ocular discomfort reduction mesured by OSDI test.

SECONDARY OUTCOMES:
Evaluate the reduction in Tear osmolarity | From enrollment to the end of treatment at 8 weeks
  Tear osmolarity test. This measurement provides important information about tear composition.
Measure the stability of the tear film | From enrollment to the end of treatment at 8 weeks
  Tear Break-Up Time (TBUT) test This measures the stability of the tear film.
Measure the tear production | From enrollment to the end of treatment at 8 weeks
  Schirmer test I (without anesthetic) at 5 minutes. This measures tear production.
Evaluate corneal staining | From enrollment to the end of treatment at 8 weeks
  Biomicroscopic observation with white light and cobalt blue light according to the Oxford scheme. It provides information on corneal health.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, available on request
URL: https://guides.lib.umich.edu/datamanagement/clinicaltrials

REFERENCES:
- [Derived] Caruso C, D'Andrea L, Rinaldi M, Senese I, Piscopo R, Costagliola C. Modified Sodium hyaluronate conjugated to riboflavin (Har(R) 0.1 %) as lubricant eyedrops in the treatment of dry eye: A prospective randomised study. Heliyon. 2024 Jul 31;10(15):e35527. doi: 10.1016/j.heliyon.2024.e35527. eCollection 2024 Aug 15. PMID 39170271